CLINICAL TRIAL: NCT05957614
Title: A Prospective Randomized Controlled Clinical Trial on the Comparison of Traditional Rehabilitation Protocol and Acupuncture-assisted Rehabilitation Protocol for Achilles Tendon Rupture
Brief Title: Effects of Acupuncture-assisted Rehabilitation Protocol for Achilles Tendon Rupture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUTHLYBLY
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: Achilles Tendon Rupture
Keywords: Rehabilitation; Acupuncture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Rehabilitation Protocol (Experimental)
  Interventions: Procedure: Traditional rehabilitation protocol
- Acupuncture-assisted Rehabilitation Protocol (Active Comparator)
  Interventions: Procedure: Acupuncture-assisted Rehabilitation Protocol

INTERVENTIONS:
Procedure: Traditional rehabilitation protocol — Rehabilitation protocol after open surgery for Achilles tendon rupture, including immobilization, early weightbearing ankle motion exercise and isolated early ankle motion exercises.
  Arms: Traditional Rehabilitation Protocol
Procedure: Acupuncture-assisted Rehabilitation Protocol — Add acupuncture treatment on the basis of traditional rehabilitation protocol.The acupuncture procedure is as follows, acupuncture treatment is carried out for half an hour every day in two weeks after surgery. The acupoints on the affected side are ST36(ZuSanLi), GB34(YangLingQuan) and SP9(YinLingQuan), and the acupoints on the healthy side are Ki3(TaiXi), bl60(KunLun) and PC7(DaLing).
  Arms: Acupuncture-assisted Rehabilitation Protocol

SUMMARY:
This prospective study is to compare the rehabilitation effect between the patients with achilles tendon rupture using traditional rehabilitation protocol and acupuncture-assisted rehabilitation protocol. The main question it aims to answer is whether acupuncture is an effective rehabilitation treatment. The patients are divided into the traditional rehabilitation group and acupuncture assisted rehabilitation group. The time of return to light sports activity and other indicators of the two groups will be compared.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical study is designed to compare the treatment outcomes of different rehabilitation protocols by dividing the patients into two groups-based on the traditional rehabilitation protocol and acupuncture-assisted rehabilitation protocol. See the text for detailed inclusion and exclusion criteria. Patients that meet all the inclusion criteria but do not meet any exclusion criteria, and who have signed the informed consent will be recruited, and each patient will be assigned a unique patient identification number, which will be used throughout the study identify the patient. All patients be treated surgically with the same suture technique. For acupuncture-assisted rehabilitation group, patients will receive additional acupuncture treatment. Investigators will collect indicators from multiple dimensions such as ankle function and pain level to compare the efficacy of the two groups.

The achilles tendon , despite being the largest and strongest tendon, is often prone to ruptures. The latest evidence48 has demonstrated that at centers using functional rehabilitation, nonoperative treatment results in similar rerupture rates but significantly lower complica- tion rates than surgical treatment. So we expect this trial to point out better rehabilitation.

In traditional Chinese acupuncture, nearly 400 acupoints on the body surface are interrelated to various functions. Acupuncture has also been widely studied for the treatment of motor system diseases. However, trials on rehabilitation of Achilles tendon rupture are still lacking.

ELIGIBILITY:
Inclusion Criteria:

* acute closed single-legged complete Achilles tendon rupture
* age of 18 to 60 years.

Exclusion Criteria:

* patients with prior Achilles tendon rupture or other situations that affected their lower limb functions or tendon healing (e.g., autoimmune disease, diabetes mellitus, systemic corticosteroid treatment).
* an inability to complete our suture technique (e.g., the distance from the rupture site to the Achilles tendon insertion was less than 3.5 cm) .
* those without rehabilitation or follow-up outcomes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The time of return to light sports activity | From operation to 1-year follow-up after the surgery
  When the patients are able to do jogging or rapid walk after the surgery, the time will be recorded.

SECONDARY OUTCOMES:
Range of motion (ROM) recovery time | From operation to 1-year follow-up after the surgery
  The recovery time will be recorded when the ROM is similar to that of the uninjured side.
Recovery time of the single-legged heel rise height (SHRH) | From operation to 1-year follow-up after the surgery
  The heel rise height is measured as the distance from the ground to the heel when the patient lift the heel while keeping the knee straight. The recovery time is noted when the SHRH is similar to that of the opposite leg.

OTHER OUTCOMES:
Visual analogue scale (VAS) | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  VAS pain score is from 0 to 10, the higher score demonstrate the more severe.
American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot score | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  The AOFAS score ranges from 0 to 100, with a healthy hindfoot receiving 100 points.
The Achilles tendon Total Rupture Score (ATRS) | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  The ATRS includes 10 items; each item has a score ranging between 0 and 10 on a Likert scale, with 100 indicating no major limitations.